CLINICAL TRIAL: NCT06261385
Title: Development of Typology-based Smoking Relapse Prevention: A Q-methodology and a Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: typology
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation
Keywords: Q-methdololgy; Relapse Prevention; Randomized Controlled Trial
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: 2-arm: Intervention group and Control group
Masking Description: open-labelled RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group, in addition to routine counselling (15-30 minutes), they will classify their identity with our screening tool (developed in Phase 2) and then apply the counselling protocol for the participants (5-10 minutes). After the counselling session, the personalized e-messages will be sent to the participants by the counsellor for 4 weeks.
  Interventions: Behavioral: typology-based intervention
- Control Group (Active Comparator): In the control group, the routine smoking cessation counselling, including generic advice on preventing smoking relapse, will be retained, and they will receive brief e-messages that only consist of general quit advice for 4 weeks.
  Interventions: Behavioral: Routine Treatment

INTERVENTIONS:
Behavioral: typology-based intervention — The typology-based intervention includes:
  1. typology-based counselling,
  2. personalized E-message based on the counselling content discussed
  3. a booklet introducing the typology of quit identity.
  All interventions and materials are delivered by smoking counselling.
  Arms: Intervention group
Behavioral: Routine Treatment — The routine smoking cessation intervention includes:
  1. Routine counselling generic advice on preventing smoking relapse
  2. Brief e-messages that consist of general quit advice for 4 weeks.
  Counsellors implement both routine practices.
  Arms: Control Group

SUMMARY:
This study aims to develop a typology-based intervention delivered by smoking cessation (SC) counselors to prevent smoking relapse in ex-smokers who recently quit. The two main research questions include (1) Can a typology-based smoking relapse prevention intervention be feasible and accepted by the smokers and SC counselors who deliver the new intervention? (2) What is the preliminary evidence on the efficacy of the typology-based smoking relapse prevention to increase tobacco abstinence in ex-smokers who have recently quit? If the intervention shows at least a small effect size (i.e. risk ratio>1.3), or the intervention is feasible while modifications can potentially increase the efficacy, a future definitive RCT is warranted.

DETAILED DESCRIPTION:
This pilot study includes three phases. The first phase will be a Q-sorting process on the Q-statements which have been developed in the pilot study. Phase 2 will be the development of a typology assessment tool, intervention protocol, and training. Phase 3 will be a pilot randomized controlled trial to examine the feasibility, acceptability and preliminary efficacy of the typology-based intervention. Ethics approval will be obtained from the Institutional Review Board of the University of Hong Kong/Hong Kong Authority Hong Kong West Cluster.

This study protocol complies with the Declaration of Helsinki and the International Conference on Harmonisation Guideline for Good Clinical Practice (ICH-GCP).

Phase 1 Q-method study (5 months) In phase 1, ex-smokers will be recruited online and in local community-based SC clinics. Mass mails including study details will be sent to all HKU staff and students. Recruitment ads will also be posted on online platforms such as Google, Facebook, and Instagram. Participants will be directed to an online Qualtrics to complete a brief screening questionnaire and provide their contact information for the sign-up process. SC clinics or services under Tung Wah Group of Hospitals, Pok Oi Hospital, Hospital Authority (HA), and Youth Quitline of the University of Hong Kong, which offer behaviour and/or pharmacological interventions. The investigators have successful experience collaborating with these service providers in recruiting smokers for several projects. For example, the investigators recruited 1,008 ex-smokers from these service providers in an HMRF-funded project in 2018-2019 (Project No. 15163001). In these clinics, potential participants shall be identified by the SC counsellors and referred to our research assistants to proceed with enrolment. In phase 3, the investigators will only recruit ex-smokers from SC clinics, because biochemical verification of both abstinence and habitual tobacco use before quitting in ex-smokers recruited from the community does not exist.

The Q-statements have been developed in our aforementioned pilot study. The Q-sorting process will be conducted on an online platform "easyHTMLQ" (Appendix 2), which is designed for completion of the Q-sorting. In this self-explanatory website, participants can easily drag the statements into the Q-sort grid according to their agreement level, and provide detailed reasons for their choices. Also, the research assistant will communicate with participants online and monitor the Q-sorting process. After the Q-sort process, the results will be documented and exported for further data analysis.

Phase 2 Intervention development (6 months) In phase 2, the investigators shall invite SC counsellors from the above SC clinics to participate in either face-to-face or online project meetings to provide feedback on the intervention protocols.

This phase aims to develop a typology assessment tool and design a typology-based intervention protocol, using the findings in Phase 1, the 3 aforementioned principles of typology-based intervention, and current smoking cessation guidelines. The screening protocol will include distinguishing statements found in Phase 1 that can characterise ex-smokers. The intervention protocol will include specific counselling principles and content for each ex-smoker class and a series of typology-based e-messages to be delivered to the corresponding class of ex-smokers via WhatsApp after counselling. The counselling shall take 5 to 10 minutes and can be fitted in current intervention protocols (5A/5R/Motivational Interview), that can address quit motivation, smoking cues and nicotine dependence.

After intervention development, the project team will invite SC counsellors for a project meeting to provide feedback on the intervention protocols. Afterwards, the project team shall revise the protocols and deliver a briefing for the SC counsellors who will deliver the intervention in Phase 3.

Phase 3 Pilot randomized control trial (7 months) The pilot 2-arm, parallel, open-labelled RCT (allocation ratio 1:1) aims to examine the feasibility, acceptability and preliminary efficacy of the typology-based intervention. SC counsellors who attend the briefing in Phase 2 will screen and recruit their SC clients to receive the typology-based intervention for smoking cessation. The SC counsellors from local clinical settings that can recruit a relatively large number of participants within the 12-week recruitment will be included, to ensure timely recruitment of sufficient participants.

During the last remote consultation with a client (mostly at 4 weeks), the SC counsellors will assess their eligibility. If they are eligible, the SC counsellors will seek their written consent and randomize them to either the intervention group or the control group. In the intervention group, in addition to routine counselling (15-30 minutes), they will classify their identity with our screening tool (developed in Phase 2) and then apply the counselling protocol for the participants (5-10 minutes). After the counselling session, the personalized e-messages will be sent to the participants by our research staff for 4 weeks.

In the control group, routine smoking cessation counselling, including generic advice on preventing smoking relapse, will be retained, and no e-messages will be sent. The investigators only deploy usual practice but not equal contact/attention treatment for the control group because the investigators aim for a superiority trial to assess the preliminary efficacy of the new intervention.

ELIGIBILITY:
Inclusion Criteria (for Ex-smoker) :

* Being a daily smoker before enrolling into the smoking cessation service
* Not using cigarettes for past 7 days
* Received at least 4 weeks of smoking cessation service before enrolling into the study
* Aged 18 years or above
* No barriers in speaking and listening Cantonese and Mandarin and reading Chinese

Exclusion Criteria (for Ex-smoker) :

* Have unstable physical or psychological conditions as advised by doctors or counsellors
* Have become pregnant in the past two months

Inclusion Criteria (for SC counsellors) :

* SC counsellors from local SC clinics under Tung Wah Group of Hospitals Integrated Center on Smoking Cessation and United Christian Nethersole Community Health Service

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
self-reported abstinence in the past 30 days at 2-month follow-up | 2 months
iScreen OFD Cotinine Saliva Test Kit (<30ng/ml) biochemical validated tobacco abstinence | 2 months
  Participants who report tobacco abstinence will be invited for a biochemical validation to test if his/her saliva cotinine is less than 30ng/ml measured by the iScreen OFD Cotinine Saliva Test Kit.
the difference of the feasibility and acceptability score of the typology-based intervention between the intervention and control group. | 2 months
  We will have 4 feasibility questions and 4 appropriateness questions for counsellor to answer from 1 (Completely disagree) to 5 (Completely agree).
  Also, we will have 4 acceptability questions for ex-smokers to answer. We would like to observe if there is a difference between the intervention group and the control group

SECONDARY OUTCOMES:
Time required for the counselling | End of all follow-up (approximately 6 month)
  The average time required for the typological counselling in minutes
Compliance rate of the SC counsellors in following the intervention protocol | End of all follow-up (approximately 6 month)
  There were 26 questions in the counselling protocol. SC counsellors have to record the number of questions asked during the typological counselling. The rate is calculated by "number of questions asked"/26.
Proportion of screened clients who participate in the RCT | End of all follow-up (approximately 6 month)
  The proportion is calculated by "Number of enrolled participants" / "Total number of participant screened"
Dropout rate of the participants who consent to the RCT | End of all follow-up (approximately 6 month)
  The dropout rate is calculated by "Number of participants dropout from study" / "Total number of enrolled participant"
Satisfaction on the SC counsellors | 2 months
  Satisfaction on the SC counsellors is measured by a 5 point Likert scale reported by the enrolled participants.
Satisfaction on the e-messages | 2 months
  Satisfaction on the e-messages is measured by a 10 point Likert scale reported by the enrolled participants.
Frequency of reading the e-messages | 2 months
  The Frequency of reading the e-messages is measured by 5 point Likert scale, which includes the option (5) I read all of them, (4) I read most of them, (3) I read half of them, (2) I read some of them, and (1) I read none of them.
Perceived effectiveness on the intervention | 2 months
  The perceived effectiveness on the intervention is measured by a 10 point likert scale. Participant will rate the usefulness of the messages in helping them to maintain smoking abstinence (10: Very useful | 0: Useless).
Satisfaction on the enrolment procedures | 2 months
  Satisfaction on the enrolment procedures is measured by a 10 point Likert scale reported by the participants (0: The enrollment procedure is slow and complicated | 10: the enrollment procedure is fast and simple).
Intention to recommend the intervention to other smokers | 2 months
  Intention to recommend the intervention to other smokers is measured by a 10 point Likert scale, 10: strongly recommended to other smokers | 0: not recommended to other smoker
Satisfaction about the intervention from SC counsellor | End of all follow-up (approximately 6 month)
  Satisfaction about the intervention from SC counsellor is measured by a 5 point Likert scale. SC counsellor will rate the effectiveness of the typological counselling in helping their client to quit smoking, from 1: very ineffective to 5: very effective.
Perceived appropriateness of the intervention length from SC counsellor | End of all follow-up (approximately 6 month)
  The perceived appropriateness of the intervention length from SC counsellor is measured by a 5 point Likert scale. SC counsellor will be asked if they agreed that the length of the typological counselling is suitable for their client, from 1 strongly disagree to 5 strongly agree.
Satisfaction on the enrolment and counselling procedures from SC counsellors | End of all follow-up (approximately 6 month)
  The satisfaction on the enrolment procedures from SC counsellors is measured by a 5 point Likert scale. Counsellors will be asked if they agreed that enrolment and counselling procedures is simple and could be easily done in the SC clinics, from 1: strongly disagree to 5: strongly agree.
Perceived effectiveness of the screening tool from SC counsellor | End of all follow-up (approximately 6 month)
  The perceived effectiveness of the screening tool from SC counsellor is measured by a 5 point Likert scale. SC counsellor will be asked if they agreed that the typological intervention can help them screen out smokers who are prone to relapse, from 1: strongly disagree to 5: strongly agree.
Perceived clients' acceptance of the intervention from SC counsellor | 2 months
  The Perceived clients' acceptance of the intervention from SC counsellor is measured by a 5 point Likert scale. Participants are asked if they agreed that counselling content provided the SC counselling gain their trust and acceptance, from 1: strongly disagree to 5: strongly agree.
Intention to apply this intervention in other clients from SC counsellors | End of all follow-up (approximately 6 month)
  Intention to apply this intervention in other clients from SC counsellors is measured by a 5 point Likert scale. SC counsellors are asked if they want to apply the typological intervention to other clients in future, 1: I will not apply it to my client in the future, 5: I want to apply it my client in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years after the completion of the relevant publications

REFERENCES:
- [Background] McGhee SM, Ho LM, Lapsley HM, Chau J, Cheung WL, Ho SY, Pow M, Lam TH, Hedley AJ. Cost of tobacco-related diseases, including passive smoking, in Hong Kong. Tob Control. 2006 Apr;15(2):125-30. doi: 10.1136/tc.2005.013292. PMID 16565461
- [Background] Census & Statistics Department (Hong Kong SAR government). Thematic Household Survey, Report No. 70: Pattern of Smoking. Hong Kong: Census & Statistics Department 2020.
- [Background] World Health Organization. A guide for tobacco users to quit. Geneva: World Health Organization; 2014.
- [Background] Lam TH. Absolute risk of tobacco deaths: one in two smokers will be killed by smoking: comment on "Smoking and all-cause mortality in older people". Arch Intern Med. 2012 Jun 11;172(11):845-6. doi: 10.1001/archinternmed.2012.1927. No abstract available. PMID 22688993
- [Background] Food and Health Bureau, Department of Health. Towards 2025: Strategy and action plan to prevent and control non-communicable diseases in Hong Kong. Hong Kong: Department of Health; 2018.
- [Background] Hartmann-Boyce J, Livingstone-Banks J, Ordonez-Mena JM, Fanshawe TR, Lindson N, Freeman SC, Sutton AJ, Theodoulou A, Aveyard P. Behavioural interventions for smoking cessation: an overview and network meta-analysis. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD013229. doi: 10.1002/14651858.CD013229.pub2. PMID 33411338
- [Background] Jackson SE, McGowan JA, Ubhi HK, Proudfoot H, Shahab L, Brown J, West R. Modelling continuous abstinence rates over time from clinical trials of pharmacological interventions for smoking cessation. Addiction. 2019 May;114(5):787-797. doi: 10.1111/add.14549. Epub 2019 Jan 29. PMID 30614586
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Background] Livingstone-Banks J, Norris E, Hartmann-Boyce J, West R, Jarvis M, Hajek P. Relapse prevention interventions for smoking cessation. Cochrane Database Syst Rev. 2019 Feb 13;2(2):CD003999. doi: 10.1002/14651858.CD003999.pub5. PMID 30758045
- [Background] Census & Statistics Department (Hong Kong SAR government). Thematic Household Survey, Report No. 64: Pattern of Smoking. Hong Kong: Census & Statistics Department 2018.
- [Background] Smith AL, Chapman S, Dunlop SM. What do we know about unassisted smoking cessation in Australia? A systematic review, 2005-2012. Tob Control. 2015 Jan;24(1):18-27. doi: 10.1136/tobaccocontrol-2013-051019. Epub 2013 Sep 11. PMID 24026163
- [Background] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159
- [Background] Luk TT, Cheung YTD, Chan HC, Fok PW, Ho KS, Sze CD, Lam TH, Wang MP. Mobile Chat Messaging for Preventing Smoking Relapse Amid the COVID-19 Pandemic: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2023 Jan 5;25(2):291-297. doi: 10.1093/ntr/ntac045. PMID 35166327
- [Background] Tajfel H, Turner JC. The Social Identity Theory of Intergroup Behavior. In: Sidanius JTJJ, editor. Political psychology: Key readings. Key readings in social psychology. New York, NY, US: Psychology Press; 2004. p. 276-93.
- [Background] Oyserman D, Smith GC, Elmore K. Identity-based motivation: Implications for health and health disparities. J Soc Iss. 2014;70(2):206-25.
- [Background] Berger J, Rand L. Shifting Signals to Help Health: Using Identity Signaling to Reduce Risky Health Behaviors. Journal of Consumer Research. 2008;35(3):509-18.
- [Background] Montes KS, Pearson MR. I am what I am: A meta-analysis of the association between substance user identities and substance use-related outcomes. Psychol Addict Behav. 2021 May;35(3):231-246. doi: 10.1037/adb0000721. Epub 2021 Apr 8. PMID 33829814
- [Background] Tombor I, Shahab L, Herbec A, Neale J, Michie S, West R. Smoker identity and its potential role in young adults' smoking behavior: A meta-ethnography. Health Psychol. 2015 Oct;34(10):992-1003. doi: 10.1037/hea0000191. Epub 2015 Jan 26. PMID 25622078
- [Background] Meijer E, Gebhardt WA, Dijkstra A, Willemsen MC, Van Laar C. Quitting smoking: The importance of non-smoker identity in predicting smoking behaviour and responses to a smoking ban. Psychol Health. 2015;30(12):1387-409. doi: 10.1080/08870446.2015.1049603. Epub 2015 Jun 3. PMID 25959600
- [Background] Susan ER, Isadore N. Q Methodology and Its Position in the Mixed-Methods Continuum. Operant Subjectivity. 2011;34(3):172-91.
- [Background] Kufeld C. A Q-Methodology study investigating the identity self-descriptions of a group of ex-smokers. England: University of Luton; 2004.
- [Background] Oyserman D. Identity-based motivation: Implications for action-readiness, procedural-readiness, and consumer behavior. J Consum Psychol. 2009;19(3):250-60.
- [Background] Watts S, Stenner P. Doing the fieldwork: participants, materials and procedure. 2012 2022/03/11. In: Doing Q Methodological Research: Theory, Method and Interpretation [Internet]. London: SAGE Publications Ltd; [69-90]. Available from: https://methods.sagepub.com/book/doing-q-methodological-research.
- [Background] Zabala A, Pascual U. Bootstrapping Q Methodology to Improve the Understanding of Human Perspectives. PLoS One. 2016 Feb 4;11(2):e0148087. doi: 10.1371/journal.pone.0148087. eCollection 2016. PMID 26845694
- [Result] GBD 2016 Risk Factors Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1345-1422. doi: 10.1016/S0140-6736(17)32366-8. PMID 28919119